CLINICAL TRIAL: NCT02652455
Title: A Pilot Clinical Trial Combining PD-1 Blockade, CD137 Agonism and Adoptive Cell Therapy for Metastatic Melanoma
Brief Title: Combining PD-1 Blockade, CD137 Agonism and Adoptive Cell Therapy for Metastatic Melanoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry); Prometheus Inc. (Industry); Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18377
Record Dates: First submitted 2016-01-08; First posted 2016-01-11 (Estimated); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Melanoma (Skin); Skin Cancer
Keywords: cutaneous; unresectable; mucosal metastatic stage III/IV melanoma
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Nivolumab; urelumab; Cyclophosphamide; fludarabine; fludarabine phosphate; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PD-1, CD137 and Adoptive Cell Therapy (Experimental): Combination Therapy and Immunotherapy as described in intervention descriptions.
  1. Nivolumab Treatment: The first 6 participants will not have pre-treatment with nivolumab and instead will be scheduled for the removal of their tumor sample for tumor Infiltrating lymphocytes (TIL) growth in the lab. The second 6 participants will receive treatment with nivolumab prior to removal of tumor sample for TIL growth; about 2 weeks after their tumor sample has been taken, these participants may receive additional infusions of nivolumab.
  2. Surgery to remove tumor for growth of TIL followed by: TIL growth process; lymphodepleting chemotherapy with cyclophosphamide and fludarabine; TIL infusion; Interleukin-2 treatment.
  Interventions: Drug: Nivolumab; Procedure: Surgery to Remove Tumor for Growth of TIL; Drug: CD137; Drug: Cyclophosphamide; Drug: Fludarabine; Biological: TIL Infusion; Drug: Interleukin-2

INTERVENTIONS:
Drug: Nivolumab — Participants entering the study after the first 6 participants only: Treatment with nivolumab prior to removal of tumor sample for TIL growth. About 2 weeks after their tumor sample has been taken, these participants may receive additional infusions of nivolumab.
  Other Names: Opdivo; PD-1 blocking antibody; BMS-936558
Procedure: Surgery to Remove Tumor for Growth of TIL — All participants: Tumor sample taken for growth of TILs. Growing the TILs takes about 4-8 weeks.
  Other Names: Tumor Infiltrating Lymphocytes (TILs); T-cell
Drug: CD137 — All participants: Anti-CD137 agonistic antibody as an agent to augment T cell proliferation in vitro. The growth of the TIL will be accelerated by the use of CD137 activating antibody in the laboratory.
  Other Names: anti-CD137 agonistic antibody; BMS-663513; 4-1BB
Drug: Cyclophosphamide — All participants: Lymphodepleting chemotherapy intravenously, beginning 3 to 6 weeks after tumor collection for TIL growth.
  Other Names: Cytoxan
Drug: Fludarabine — All participants: Lymphodepleting chemotherapy intravenously, beginning after first 2 days of cyclophosphamide.
  Other Names: Fludara
Biological: TIL Infusion — After completing one week of lymphodepleting chemotherapy, all participants will be admitted back into the hospital for IV infusion of the TIL cells.
Drug: Interleukin-2 — After TIL infusion, in-patient high dose IL-2 treatment.
  Other Names: IL-2; Proleukin; Aldesleukin

SUMMARY:
The purpose of this Pilot Study is to investigate the safety, side effects, and benefits of tumor- infiltrating lymphocytes (TILs) when they are given with the drug nivolumab. Nivolumab is a type of immunotherapy - a drug that is used to boost the ability of the immune system to fight cancer, infection, and other diseases.

The primary endpoints of this pilot trial will be the safety and feasibility of the treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* Must have unresectable cutaneous or mucosal metastatic stage III/IV melanoma, and in the opinion of the institutional principal investigator (PI) is an acceptable candidate for adoptive cell therapy (ACT) with high dose IL-2.
* Must have anticipated residual measurable disease after resection of target lesion(s) for TIL growth.
* Patients who have been previously treated for metastatic melanoma may be included (e.g., prior treatment with Rapidly Accelerated Fibrosarcoma (BRAF) inhibitors and/or ipilimumab will be allowed), provided that they have had a three week 'washout' prior to signing consent and have not been treated with a Programmed Death-1 (PD-1) blocking antibody.
* Age greater than or equal to 18 years.
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 - 1.
* Women of childbearing potential must have a negative serum pregnancy test within seven days of screening and within 24 hours prior to the start of each nivolumab dose.
* Adequate renal, hepatic and hematologic function.
* Patients must have a positive screening Epstein Barr Virus (EBV) antibody titer on screening test as this is required to protect against EBV infection during the time of lymphodepletion.
* Patients with antibiotic allergies per se are not excluded; although the production of TIL for adoptive transfer includes antibiotics, extensive washing after harvest will minimize systemic exposure to antibiotics.
* At screening, patients with ≤ 3 untreated central nervous system (CNS) metastases may be included provided none of the untreated lesions are > 1 cm in greatest dimension, and there is no peri-tumoral edema present on brain imaging (MRI or CT if MRI is contraindicated), and if the patients with CNS metastases are not taking prednisone >10 mg or equivalent daily.
* At screening, patients with ≤ 3 CNS metastases and each ≤ 1 cm size that were treated with either surgical resection and/or radiation therapy may be included. Patients may be included if the largest lesion is ≤ 1 cm, and there is no evidence of progressive CNS disease on brain imaging at least 30 days after definitive treatment, and if the patients with CNS metastases are not taking prednisone >10 mg or equivalent daily.
* At screening, patients with> 1 cm or > 3 in number treated CNS metastases may be included if there is no evidence of progressive CNS disease on brain imaging at least 90 days after treatment with surgery and/or radiation therapy, and if the patients with CNS metastases are not taking prednisone >10 mg or equivalent daily.

Exclusion Criteria:

* Patients with active systemic infections requiring intravenous antibiotics, coagulation disorders, or other major medical illness of the cardiovascular, respiratory or immune system, which in the opinion of the PI or treating co-investigator is not acceptable risk for ACT, are excluded.
* Patients who have received prior immunotherapy whose side effects have resulted in a requirement of immunosuppressive medications (>10 mg of prednisone daily or equivalent daily steroid daily, or infliximab, cyclosporine or equivalent immunosuppressive medication) or who have other autoimmune conditions that require immunosuppressive medications as above at the time of screening are excluded.
* Patients who test positive for Human Immunodeficiency Virus (HIV), Hepatitis B surface antigen, Hepatitis B core antibody, Hepatitis C antibody, Human T-lymphotropic Virus (HTLV) I or II antibody, or are both Rapid plasma reagin (RPR) and Fluorescent treponemal antibody (FTA) positive are excluded.
* Patients who are pregnant or nursing are excluded.
* Patients with a significant psychiatric disease, who in the opinion of the principal investigator or his designee, would prevent adequate informed consent or render immunotherapy unsafe will be excluded.
* Patients with > 3 untreated CNS metastases or evidence of peri-tumoral edema will be excluded, or patients with CNS metastases of any status who are taking prednisone >10 mg or equivalent steroid daily will be excluded.
* Patients with ≤ 3 untreated CNS metastases but with at least one lesion >1 cm or peri-tumoral edema will be excluded, or patients with CNS metastases of any status who are taking prednisone >10 mg or equivalent steroid daily will be excluded.
* Patients with invasive malignancy other than melanoma at the time of enrollment and within 2 years of screening are excluded, except for: adequately treated (i.e. with curative intent) basal or squamous cell carcinoma, in situ carcinoma of the cervix, in situ ductal adenocarcinoma of the breast, in situ prostate cancer, or limited stage bladder cancer or other any other cancers from which the patient has been disease-free for at least 2 years.
* Patients with treated CNS metastases > 1 cm or > 3 in number will be excluded if there is evidence of progressive CNS disease on brain imaging at least 90 days after treatment with surgery and/or radiation therapy, or patients with CNS metastases of any status who are taking prednisone >10 mg or equivalent will be excluded.
* Male patients with female partners of childbearing potential who do not agree to use two FDA-accepted forms of contraception during sexual intercourse with women of child-bearing potential from the start of PD-1 antibody therapy and up to at least 31 weeks from the last dose of nivolumab are excluded.
* Females of childbearing potential who do not agree to use 2 FDA forms of contraception according to study guidelines
* Prior systemic therapy with a PD-1 blocking antibody
* Patients who are greater than age 50, or who have a history of coronary artery disease, will be required to undergo cardiac stress testing within 6 months of screening and will be excluded if there is evidence of reversible ischemia.
* Patients who have a significant history of pulmonary disease that necessitates the use of supplemental oxygen, is associated with dyspnea on walking one block or less, or requires inhaler therapy more than once per week will be required to undergo pulmonary function testing within 6 months of screening and will be excluded if forced expiratory volume 1 (FEV1), forced vital capacity (FVC), or diffusion lung capacity for carbon monoxide (DLCO) is less than 65% of predicted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of Study Related Adverse Events | Up to 27 months
  Safety will be determined by assessing toxicity based upon Common Terminology Criteria for Adverse Events (CTCAE) v4.

CONTACTS AND LOCATIONS:
Overall Officials: Amod Sarnaik, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/